CLINICAL TRIAL: NCT05445180
Title: Investigating the Neural Correlates of Cognitive Function Associated With Cannabis Abstinence in Psychosis Patients and Non-Psychiatric Controls With Cannabis Use
Brief Title: Investigating the Neural Correlates of Cognitive Function in Psychosis Patients and Non-Psychiatric Controls With Cannabis Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, Rachel Rabin, Assistant Professor, Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IUSMD-21-11
Record Dates: First submitted 2022-05-18; First posted 2022-07-06 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Psychotic Disorders; Cannabis Use Disorder; Cannabis Dependence; Cannabis Use; Schizophrenia; Psychosis; Cognitive Dysfunction; Memory Impairment; Neuroimaging
MeSH Terms: conditions — Psychotic Disorders; Marijuana Abuse; Schizophrenia; Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research Assistant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Psychosis patients with cannabis use (Abstinent) (Experimental): Psychosis patients with cannabis use will receive contingency management to encourage cannabis abstinence for 28 days
  Interventions: Behavioral: Contingency management
- Psychosis patients with cannabis use (Non-abstinent) (No Intervention): Psychosis Patients with cannabis use who will continue to use cannabis as usual
- Non-Psychiatric controls with cannabis use (Abstinent) (Experimental): Non-Psychiatric controls with cannabis use will receive contingency management to encourage cannabis abstinence for 28 days
  Interventions: Behavioral: Contingency management
- Non-Psychiatric controls with cannabis use (Non-abstinent) (No Intervention): Non-Psychiatric Controls with cannabis use will continue to use cannabis as usual
- Non-Psychiatric Controls without cannabis use (No Intervention): Non-Psychiatric controls without cannabis use

INTERVENTIONS:
Behavioral: Contingency management — Contingency management will be used to encourage abstinence
  Arms: Non-Psychiatric controls with cannabis use (Abstinent); Psychosis patients with cannabis use (Abstinent)

SUMMARY:
Cognitive impairment is well established in people with psychosis and is associated with cannabis use. The current study will investigate the neurobiological basis of cognitive change associated with 28-days of cannabis abstinence in people with psychosis and non-psychiatric controls with cannabis use. Participants will be randomized to a cannabis abstinent group or a non-abstinent control group and will undergo magnetic resonance imaging at baseline and following 28-days of abstinence. This study will help characterize the neuropathophysiological processes underlying cognitive dysfunction associated with cannabis use and its recovery which may guide the development of novel interventions for problematic cannabis use.

DETAILED DESCRIPTION:
Background/Importance: Cognitive impairment is well established in people with psychosis and is associated with cannabis use. Despite high rates of cannabis use among people with psychosis and the general population, cannabis' effects on cognition and the brain and their recovery remain unclear. Therefore, this study will investigate the neurobiological basis of changes in cognitive processes associated with cannabis abstinence in people with psychosis and non-psychiatric controls.

Aims: To examine the effects of 28-days of cannabis abstinence in psychosis patients with cannabis use and non-psychiatric controls with cannabis use on (i) brain activity (paired with a memory task); (ii) brain morphology; (iii) to determine if changes in memory following 28-days of abstinence correlate with changes in brain activity and/or morphology and (iv) to determine if baseline brain function and morphology can predict successful abstinence.

Methods: Seventy-four psychosis patients with cannabis use and 60 non-psychiatric controls with cannabis use will be randomized to: (1) contingency reinforcement where biochemically verified abstinence at day 28 will be rewarded; or (2) a non-abstinent control group. The investigators will also recruit a group of healthy non-psychiatric controls (n=40) to determine if neural outcomes in cannabis-using participants do indeed normalize ("recover") following abstinence. Participants will undergo structural and functional magnetic resonance imaging while completing a memory task at baseline (pre-abstinence) and following 28-days of abstinence. Urine samples will be collected twice weekly for abstinence verification.

Relevance: This study will help to characterize the neuropathophysiological processes underlying cognitive dysfunction associated with cannabis use in people with psychosis and non-psychiatric controls which may help to guide the development of novel neurobiologically-informed interventions to treat problematic cannabis use.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent in English or French
* Heavy cannabis use (defined as weekly cannabis use for at six months) and/or DSM-5 diagnosis of CUD
* Have a Full-Scale IQ ≥ 75
* Meet DSM-5 criteria for a psychotic disorder (psychosis patient arm only)
* Be an outpatient receiving a stable dose of medication(s) for at least two months (psychosis patient arm only)
* Clinically stable (as measured by the PANSS-6, total score <30) (psychosis patient arm only)

Exclusion Criteria:

* current SUD (other than CUD)
* MRI contraindications
* Positive urine screen for psychoactive substances other than cannabis, nicotine, or caffeine
* Current suicidal or homicidal ideation
* Head injury requiring hospitalization or loss of consciousness > 5 minutes
* Current medical diseases that requires hospitalization or regular monitoring
* Being pregnant
* DSM-5 Axis 1 diagnosis (other than CUD) (non-psychiatric controls only)
* Taking psychotropic medication

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in fMRI brain activity pattern | Baseline, Day 28
  fMRI will be used to measure differences between baseline (day 0) and day 28 in hemodynamic (BOLD) responses while participants complete a memory task
Change in behavior during fMRI task | Baseline, Day 28
  Behavioral responses (episodic memory performance) will be recorded by an external button box. These responses will be used to assess encoding accuracy during an episodic memory task.

SECONDARY OUTCOMES:
Change in brain morphology: gray matter volume | Baseline, Day 28
  Using MRI, changes in gray matter volume will be analyzed from baseline (day 0) to day 28
Change in brain morphology: cortical thickness | Baseline, Day 28
  Using MRI, changes in cortical thickness will be analyzed from baseline (day 0) to day 28
Change in brain morphology: diffusion | Baseline, Day 28
  Using MRI, changes in diffusion based measures will be analyzed from baseline (day 0) to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Rabin, Ph. D., Principal Investigator — Douglas Mental Health University Institute
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Contact the P.I.
Supporting Information: Study Protocol, SAP, Analytic Code
Access Criteria: Contact the P.I.